CLINICAL TRIAL: NCT03496116
Title: The Influence of Electronic Cigarette Heater Resistance on Nicotine Delivery, Heart Rate, Subjective Effects and Puff Topography
Brief Title: The Influence of Electronic (ECIG) Heater Resistance on ECIG Acute Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20012671
Record Dates: First submitted 2018-04-02; First posted 2018-04-12 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ECIG Session: 0.5 Ohms, 3 mg (Experimental): Heating coil resistance 0.5 Ohms Liquid nicotine concentration 3 mg
  Interventions: Other: ECIG Session
- ECIG Session 0.5 Ohms, 8 mg (Experimental): Heating coil resistance 0.5 Ohms Liquid nicotine concentration 8 mg
  Interventions: Other: ECIG Session
- ECIG Session 1.5 Ohms, 3 mg (Experimental): Heating coil resistance 1.5 Ohms Liquid nicotine concentration 3 mg
  Interventions: Other: ECIG Session
- ECIG Session 1.5 Ohms, 8 mg (Experimental): Heating coil resistance 1.5 Ohms Liquid nicotine concentration 8 mg
  Interventions: Other: ECIG Session

INTERVENTIONS:
Other: ECIG Session — Participants will complete four sessions using an e-cigarette, including a 10-puff product use bout followed by a 60-minute ad lib bout over an approximately 4-hour period. The study conditions for each session (i.e., heater resistance and nicotine combinations) will be Latin-square ordered.

SUMMARY:
The purpose of this study is to measure the individual and combined influence of electronic cigarette (ECIG) heating element resistance and liquid nicotine concentration on ECIG acute effects. Thirty-two experienced ECIG users will complete four independent laboratory sessions that will differ by heater resistance (0.5 ohm or 1.5 ohm) and liquid nicotine concentration (3 or 8 mg/ml). Other factors such as voltage, liquid solvent ratio, and liquid flavor will be held constant. Plasma nicotine concentration, subjective effects, and puffing behavior will be recorded for each condition.

DETAILED DESCRIPTION:
Electronic cigarettes (ECIGs) are a popular and rapidly evolving class of products. ECIG users can manipulate several device features including liquid nicotine concentration (mg/ml) and heating element resistance (ohms). An emerging class of ECIG models includes "sub-Ohm" devices that employ low resistance heaters that are often used to achieve high device power. Some clinical laboratory data suggest that high power devices deliver nicotine to the user effectively, even when paired with a low liquid nicotine concentration. However, given that ECIG heater resistance and liquid nicotine concentration have not been manipulated in clinical laboratory studies, the influence of these factors on ECIG acute effects remain unclear. The purpose of this clinical laboratory study is to measure the influence of heater resistance and liquid nicotine concentration on ECIG acute effects. Participants will attend the lab for four experimental sessions where they use an ECIG. For each session, the participants will be randomly assigned (like the flip of a coin) to receive an ECIG with one of two different levels of heating coil resistance (which will determine overall device power) and one of two different liquid nicotine concentrations. The four sessions will begin at approximately the same time each day, will be separated by at least 48 hours, and will not occur more than two times per week. The primary hypotheses are that the low resistance heater paired with the 8 mg/ml liquid nicotine concentration, will result in greater nicotine delivery and subjective effect profiles, suggestive of higher abuse potential. Results from this study will further our understanding of the factors that influence the dependence potential of ECIGs and could inform future regulation of these devices.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent, attend the lab and abstain from nicotine/tobacco as required, and use designated products according to study protocol
* Experienced ECIG users (use ≥1 ml of ECIG solution daily, use ECIG solution with a nicotine concentration ≥3 mg/ml, and have used their ECIG for ≥3 months)
* Urine cotinine test result ≥ 3

Exclusion Criteria:

* History of organ-related diseases or current psychiatric condition
* Regular use of prescription medication other than vitamins or birth control
* Past month use of cocaine, opioids, benzodiazepines, or methamphetamine
* Using marijuana greater than 10 days in the past 30 and/or alcohol greater than 25 days in the past 30 days
* Pregnant or breastfeeding women
* Weight less than 110 pounds
* Daily use of >5 cigarettes or use of other tobacco products (i.e., hookah, cigars) >3 times a week

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Cmax: Plasma nicotine concentration (ng/ml) | Six blood samples are collected at each of the 4 visits. During each session, blood samples are collected 90,100,160,185,205,225 minutes into the session which lasts approximately 4 hours.

SECONDARY OUTCOMES:
Withdrawal suppression: Hughes-Hatsukami Withdrawal Scale | Collected six times at each of the 4 visits. During each session, questions are collected 90,100,160,185,205,225 minutes into the session which lasts approximately 4 hours.
  Contains 11 items. Administered on a computerized visual analogue scale that consists of a phrase centered on a horizontal line with "not at all" on the left and "extremely" on the right.. Responses range from 0-100.
Withdrawal suppression: Direct effects of nicotine scale | Collected six times at each of the 4 visits. During each session, questions are collected 90,100,160,185,205,225 minutes into the session which lasts approximately 4 hours.
  Contains 9-items. Administered on a computerized visual analogue scale that consists of a phrase centered on a horizontal line with "not at all" on the left and "extremely" on the right.. Responses range from 0-100.
Withdrawal suppression: Tiffany Drobes Questionnaire of Smoking Urges | Collected six times at each of the 4 visits. During each session, questions are collected 90,100,160,185,205,225 minutes into the session which lasts approximately 4 hours.
  Contains 10 items. Participants will be asked to rate each phrase on a 7-point scale ranging from 0 (Strongly disagree) to 7 (Strongly agree). The items from this scale will form two factors: Factor 1 (intention to smoke) and Factor 2 (anticipation of relief from abstinence symptoms).
Withdrawal suppression: Direct effects of ECIG use scale | Collected six times at each of the 4 visits. During each session, questions are collected 90,100,160,185,205,225 minutes into the session which lasts approximately 4 hours.
  Contains 14-items. Administered on a computerized visual analogue scale that consists of a phrase centered on a horizontal line with "not at all" on the left and "extremely" on the right. Responses range from 0-100.
Other subjective effects: General Labeled Magnitude Scale | Collected six times at each of the 4 visits. During each session, questions are collected 90,100,160,185,205,225 minutes into the session which lasts approximately 4 hours.
  Contains 4-items. This category-ratio scale contains seven semantic labels that increase in sensitivity including: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable sensation of any kind." Responses will be coded on a 0-100 scale.
Other subjective effects: Labeled Hedonic Scale | Collected six times at each of the 4 visits. During each session, questions are collected 90,100,160,185,205,225 minutes into the session which lasts approximately 4 hours.
  Contains 4-items. This category-ratio scale contains ten semantic labels, intended to assess participant liking or disliking of sensations experienced in the general labeled magnitude scale.. Semantic labels include: "most liked sensation imaginable", "like extremely", "like very much", "like moderately", "like slightly", "dislike slightly", "dislike moderately", "dislike very much", "dislike extremely" and "most disliked sensation imaginable". Responses will be coded on a 0-100 scale.
Puff Topography: puff duration | Collected twice at each of the 4 visits. During each session, puff duration is measured at 95 and 225 minutes.
  Puff duration is the measurement of the length of participant puffs in seconds during a 10-puff directed puffing bout (lasting 5-minutes) and during the 60-minute ad libitum bout where participants are instructed to puff as much or as little as they like on the ECIG.
Puff Topography: puff volume | Collected twice at each of the 4 visits. During each session, puff duration is measured at 95 and 225 minutes.
  Puff volume is the measurement of the size of participant puffs in milliliters during a 10-puff directed puffing bout (lasting 5-minutes) and during the 60-minute ad libitum bout where participants are instructed to puff as much or as little as they like on the ECIG.
Puff Topography: puff velocity | Collected twice at each of the 4 visits. During each session, puff duration is measured at 95 and 225 minutes.
  Puff velocity is the measurement of the speed of participant puffs in milliliters per second during a 10-puff directed puffing bout (lasting 5-minutes) and during the 60-minute ad libitum bout where participants are instructed to puff as much or as little as they like on the ECIG.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Eissenberg, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided